CLINICAL TRIAL: NCT07069387
Title: Comprehensive Digital Adherence and Remote Engagement to Optimise Treatment Adherence for Tuberculosis Patients (CARE-TB Study) in Selangor, Malaysia: An Effectiveness-Implementation Science Study
Brief Title: Pharmacist-led Digital Interventions to Improve Tuberculosis Treatment Adherence
Acronym: CARE-TB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NMRR ID 23-03504-DLE (IIR)
Record Dates: First submitted 2025-06-12; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-04

CONDITIONS: Tuberculosis (TB)
Keywords: tuberculosis; active tuberculosis; monitoring; video observed therapy; education; pharmacist; digital; implementation science; cost; motivational
MeSH Terms: conditions — Tuberculosis; Latent Tuberculosis | interventions — Motivational Interviewing; Counseling; Educational Status; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care arm (Active Comparator): Directly observed therapy (healthcare or caretaker-based)
  Interventions: Behavioral: Standard Care
- CARE-TB arm (Experimental): CARE-TB package includes pharmacist-led asynchronous video observed therapy, digital medication reminders, telecounselling and e-learning for patients.
  Interventions: Behavioral: CARE-TB digital adherence package

INTERVENTIONS:
Behavioral: CARE-TB digital adherence package — CARE-TB package includes pharmacist-led asynchronous video observed therapy, digital medication reminders, telecounselling and e-learning for patients.
  Other Names: video observed therapy; motivational interviewing; counselling; education; reminder; digital intervention
  Arms: CARE-TB arm
Behavioral: Standard Care — Directly observed therapy at any government healthcare facility (by nurses) or at home (by caretaker)
  Other Names: Directly observed therapy; In-person dose monitoring
  Arms: Standard care arm

SUMMARY:
The gold standard for tuberculosis (TB) treatment support requires directly observed therapy (DOT), which means a trained health worker observes the patient swallow each dose of medication every day for 2 months. Despite the practice of DOT in Malaysia, 1 in 20 patients are loss-to-follow-up and non-adherent to treatment. Sub-optimal adherence due to poor treatment acceptability and social desirability promotes TB treatment failure, disease relapse, on-going transmission, drug resistance, and death. Telemedicine offers a flexible and less invasive option to support TB treatment adherence. Despite 97% internet and smartphone penetration rates, the practical implementation of digital adherence strategies to support and monitor TB treatment remains untested in Malaysia. The investigators propose to design, implement, and measure the effectiveness of a comprehensive, pharmacist-led digital solution for TB treatment support called CARE-TB which combines a package of asynchronous video-observed therapy, digital reminders, telecounselling and e-learning. In this multi-method effectiveness-implementation (Type 2) study using the Exploration, Preparation, Implementation and Sustainment (EPIS) framework, the investigators aim 1) To identify patient and provider-level facilitators and barriers to CARE-TB adoption via qualitative evaluation and to design a stakeholder-informed implementation strategy, (2) To assess effectiveness of CARE-TB strategy by evaluating (i) implementation outcomes, (ii) patient health outcomes, and (iii) service outcomes, and (3) To evaluate the cost-effectiveness of CARE-TB compared to standard of care from a societal perspective. This study will leverage digital platforms to expand the reach of TB adherence support, enhance adherence to TB treatment and improve treatment completion rates, while utilising existing personnel and resources in among the busiest TB treatment centres in the country.

ELIGIBILITY:
Inclusion Criteria:

1. Microbiologically confirmed pulmonary TB (smear- or culture-positive PTB)
2. 18 years old or older
3. Able to give consent and physically able to participate in the study
4. Own a video-recording device with internet connectivity
5. Within the first 3 weeks of intensive phase TB treatment

Exclusion Criteria:

1. Complicated TB disease including TB meningitis, TB bone/joint, and disseminated TB with planned treatment duration of 9 to 12 months.
2. Confirmed or suspected drug-resistant (DR)-TB
3. Documented cognitive, motor, or visual disability that will hinder video device use and lack assistance of a caretaker
4. Receiving injectable anti-TB drugs
5. Incarceration or other involuntary detention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Medication adherence (Binary outcome) | 8 weeks following enrollment
  Completed ≥ 80% scheduled observations during the 8 weeks following enrolment.

SECONDARY OUTCOMES:
Adherence rate (Continuous outcome) | 8 weeks following enrolment
  Proportion of doses observed over 8 weeks (Dose observed divided by total observable doses prescribed)
Proportion of TB treatment completion, death, loss to follow up, and hospitalization | From enrolment till 6 months or treatment completion/ termination
  Proportion of patients completing TB treatment, died, are lost to follow-up or hospitalized during TB treatment
TB cure rate | At 6 months of treatment
  Proportion of microbiological TB clearance (e.g. AFB smear/ MTB PCR/ MTB culture)
Adverse event reporting | From enrolment till 6 months of treatment
  Number of adverse events or adverse drug reactions reported during TB treatment
EQ-5D-5L Health-related Quality of Life (HRQoL) | At baseline, 2 months and 6 months of treatment
  HRQoL will be assessed using the EuroQol 5-Dimension 5-Level (EQ-5D-5L) questionnaire.
  Unit of Measure: EQ-5D index score (range: -0.281 to 1.000 based on country-specific value set)
  Interpretation: Higher scores indicate better health-related quality of life.
SF-12 Health-related Quality of Life (HRQoL) | At baseline and 2 months of treatment
  The 12-Item Short Form Survey (SF-12) will be used to assess participants' health-related quality of life. Two summary scores will be generated: the Physical Component Summary (PCS) and the Mental Component Summary (MCS).
  The scoring scale is from 0 to 100, the higher the score the better the health related quality of life.
Implementation Outcomes: Acceptability, Feasibility, Appropriateness (Quantitative measure) | At 2 months and 6 months of treatment
  Implementation outcomes will be assessed using the combined Acceptability of Intervention Measure (AIM), Feasibility of Intervention Measure (FIM), and Intervention Appropriateness Measure (IAM) questionnaire.
  Unit of Measure: Total and individual mean scores on 5-point Likert scale (1 = completely disagree, 5 = completely agree)
  Scoring: Each subscale consists of 4 items; subscale scores range from 4 to 20
  Interpretation: Higher scores indicate greater perceived acceptability, feasibility, or appropriateness of the intervention
Perceived acceptability, feasibility, and fit of the intervention (Qualitative measure) | After 6 months of implementation phase
  Semi-structured qualitative interviews and focus group discussions will explore participants' perceptions of the intervention's acceptability, feasibility, and fit.
  Unit of Measure: Thematic findings from qualitative analysis
  Interpretation: Interview data will be thematically coded and analyzed to identify key barriers, facilitators, and contextual factors.
Adoption rate | Through study completion, an average of 1 year
  Rate of uptake (number of participants who agree to use the CARE TB strategy divided by total number offered)
Patient fidelity to intervention | 8 weeks following enrolment
  Rate of drop-out (count of individuals who fulfill any of the following: withdraw from the study, switch arms, appointment no-show)
Healthcare providers (HCP) fidelity to intervention | 8 weeks following enrolment
  Rate of reengagement attempt (count of reminders sent to reestablish VOT over total number of missed VOT appointments)

CONTACTS AND LOCATIONS:
Overall Officials: Reena Rajasuriar, Principal Investigator — University of Malaya
Locations (1):
- Sungai Buloh Hospital, Sungai Buloh, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported following deidentification.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Beginning 3 months following publication and no end date.
Access Criteria: Investigators whose proposed used of data has been approved by independent review. Proposals should be submitted to kohhuimoon@moh.gov.my. To gain access, a data sharing agreement must be signed.